CLINICAL TRIAL: NCT00168441
Title: A Study Evaluating Botulinum Toxin Type A in Subjects With Postherpetic Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-066
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A

SUMMARY:
4-month study including a 30-day baseline phase

ELIGIBILITY:
Inclusion Criteria:

* Postherpetic neuralgia for more than 3 months after the healing of a herpes zoster skin rash.

Exclusion Criteria:

* Previous use of botulinum toxin of any serotype or immunization to any botulinum toxin serotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Pain score

SECONDARY OUTCOMES:
Various Quality of Life questionnaires
Reduction in area of pain/allodynia